CLINICAL TRIAL: NCT00319852
Title: Immunogenicity and Safety of Tetraxim Versus Local DTP + IPV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2I28
Record Dates: First submitted 2006-04-28; First posted 2006-04-27 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Pertussis; Diphtheria; Poliomyelitis; Tetanus
Keywords: Diphteria;; Tetanus;; Pertussis;; Poliomyelitis;; acellular
MeSH Terms: conditions — Whooping Cough; Diphtheria; Poliomyelitis; Tetanus | interventions — Tetanus Toxoid; Diphtheria-Tetanus-acellular Pertussis Vaccines

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: DTaP-IPV combined vaccine
- 2 (Active Comparator)
  Interventions: Biological: DTaP vaccine

INTERVENTIONS:
Biological: DTaP-IPV combined vaccine — 0.5 mL, IM
  Other Names: TETRAXIM™: Diphtheria, Tetanus, Polio, Acellular Pertussis
  Arms: 1
Biological: DTaP vaccine — 0.5 mL, IM
  Other Names: DTaP vaccine (CJ purified PDT vaccine ™)
  Arms: 2

SUMMARY:
The present clinical study will assess the immunogenicity and reactogenicity of Sanofi Pasteur's DTaP-IPV combined vaccines as a three-dose primary vaccination at 2, 4 and 6 months of age compared to commercially available vaccines in order to meet the requirements for registration of the product in South Korea.

Primary objective To demonstrate the non-inferiority in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3) and seroconversion/vaccine response rates to Pertussis antigens (PT, FHA) of Sanofi Pasteur's DTaP-IPV combined vaccine versus commercially available Biken's DTaP (CJ purified PDT vaccine ™) and Aventis Pasteur's IPV (IMOVAX POLIO) monovalent vaccines, one month after the three-dose primary vaccination.

Secondary objectives

1. Immunogenicity: To assess the non-inferiority in terms of seroprotection rates (Diphtheria, Tetanus, Polio types 1, 2 and 3) and seroconversion / vaccine response rates to Pertussis antigens (PT, FHA) of Sanofi Pasteur's DTaP-IPV combined vaccine versus historical reference (Study E2I03294 - France). To assess and describe the immunogenicity of the study vaccines in both groups.
2. Safety: To assess and describe the safety of the study vaccines after each dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 56 to 70 days inclusive on the day of inclusion
* Born at full term pregnancy (>37 weeks) with a birth weight ≥ 2.5 kg
* Informed consent form signed by the parent(s) or other legal representative
* Able to attend all scheduled visits and to comply with all trial procedures

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period.
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as long-term systemic corticosteroids therapy.
* Systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past or planned administration during the trial (including immunoglobulins).
* Any vaccination in the 3 weeks preceding the first trial vaccination.
* History of diphtheria, tetanus, pertussis, poliomyelitis infection (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases with the trial vaccine or another vaccine.
* Thrombocytopenia or a bleeding disorders contraindicating intramuscular vaccination
* History of major neurological diseases or seizures.
* Febrile illness (rectal temperature ≥ 38.0°C or axillary temperature ≥ 37.4°C) on the day of inclusion.
* Known family history of congenital or genetic immuno-deficiency.

Ages: 56 Days to 70 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 442 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of Sanofi Pasteur's DTaP-IPV combined vaccine versus commercially available Biken's DTaP and Aventis Pasteur's IPV (IMOVAX POLIO) monovalent vaccines. | 1 month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com